CLINICAL TRIAL: NCT00224250
Title: Ultrasonographic Assessment of the Uterine Scarring Process Following Closure of the Uterus in One Versus Two Layer Technique.
Brief Title: Ultrasound Study of the Uterine Healing Process After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 27269
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Myometrial Remodeling

INTERVENTIONS:
Procedure: One- versus two-layer hysterotomy closure

SUMMARY:
Our hypothesis is that there is no difference in the healing process in those women who have a one- or two-layer uterine closure at the time of cesarean delivery.

DETAILED DESCRIPTION:
We are recruiting women who are presenting for their first (primary) cesarean delivery. They will be randomized to one- or two-layer myometrial closure at the time of their cesarean delivery. Ultrasound will be used to serially assess the myometrial thickness and myometrial remodeling process.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* term pregnancy
* Kerr uterine incision employed
* age > 18

Exclusion Criteria:

* Pain score > 4
* Current cesarean delivery for non-reassuring fetal status or other emergent situation (eg. maternal bleeding, etc.)
* Prior cesarean section
* Prior uterine surgery
* Hysterotomy other than Kerr (low transverse) incision in current cesarean
* Extension of the uterine incision in current cesarean
* Multifetal pregnancy
* Maternal diabetes mellitus
* Maternal connective tissue disorder
* Uterine malformation
* Uterine myomas (fibroids) in the anterior lower uterine segment
* Chorioamnionitis
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-01

PRIMARY OUTCOMES:
myometrial thickness

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hamar, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Hamar BD, Saber SB, Cackovic M, Magloire LK, Pettker CM, Abdel-Razeq SS, Rosenberg VA, Buhimschi IA, Buhimschi CS. Ultrasound evaluation of the uterine scar after cesarean delivery: a randomized controlled trial of one- and two-layer closure. Obstet Gynecol. 2007 Oct;110(4):808-13. doi: 10.1097/01.AOG.0000284628.29796.80. PMID 17906013